CLINICAL TRIAL: NCT01989715
Title: Body Posture Assessment Considering Jaws Position Before and After Orthognathic Surgery on Adult Patient.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-A00634-41; 2013-15 (Other: AP HM)
Record Dates: First submitted 2013-09-25; First posted 2013-11-21 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Orthognathic Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- adult patients waiting for orthognathic surgery (Experimental)
  Interventions: Other: analyzing the position of the body, muscle activity

INTERVENTIONS:
Other: analyzing the position of the body, muscle activity

SUMMARY:
Postural balance on both feet, characteristic of the human species, is possible by the tension of muscle of the whole body from toes to head.

Body position depends on many inputs such as vision, vestibule, skin receptors, states of muscle tension receptors. Information is integrated in a complex nervous system via the ascending and descending pathways. The information is then analyzed to provide feedback on body position. Any variation of body position, induces a variation of the center of pressure. Impaired body positioncan cause pain (back pain, neck pain) or long-term deformation (including scoliosis or kyphosis).

Maxillas position, via the activity of masseter and temporal muscles, acts on the muscle chain that controls posture. Incorrect positioning of the jaw in the three directions of space seems to create an asymmetric masticatory muscles activity and thus destabilize the muscle chain responsible for body position. Repositioning maxillas by orthognathic surgery could alter the body posture via changing the activity of the masticatory muscles.

However, nowadays no clear link has been demonstrated between maxillas repositioning and body posture modification.

The purpose of this study is to highlight the link between posture and jaws position, by analyzing the variation of the masticatory muscles activity and, the changes in body center of pressure before and after orthognathic surgery of jaws standardization.

In this study each patient will be evaluated in terms of occlusion and body posture before surgery and after surgery (2 months) by the same protocol. The surgery will be performed in the Maxillofacial Surgery service - Pr BLANC and assessment will take place in the dentistry department - Prof. Salvadori La Timone Hospital, Marseille.

The assessment includes the body posture study with a stabilometric platform (eyes open / eyes closed and with / without tooth contact), and analysis of the head orientation relative to the vertical. Electromyographic muscle masseter assessment (jaw with/without contact ) are devoted to check the evolution of the developed forces, and hand strength will be recorded using a dynamometer.

All these data will be recorded for all the patients. Patients will be divided into four subgroups: (1) maxillary endognathia, (2) mandibular prognathism , (3) mandibular retrognathia and (4 mandible repositioning.

Statistical analysis is aimed at validating or not the hypothesis of changes in body posture caused by surgical maxillas repositioning.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 to 60 years)
* patients waiting for orthognathic surgery

Exclusion Criteria:

* Patient prone to vertigo, dizziness, loss of understanding are, accouphènes.
* Patient with acute pain of migraine-type neck pain, back pain, arthritis, tendonitis.
* Patient with oral pain (acute periodontitis, caries, abscesses)
* Patient with orthopedic prosthesis.
* Patient on muscle relaxant treatment, tranquilizer, antidepressant
* Patient over 60 years of age.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-11 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
postural assessment | 6 mois
  Analysis before and after orthognathic surgery

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France